CLINICAL TRIAL: NCT03487445
Title: A Multi-center, Open-label, Randomized, Study to Assess the Onset of Platelet Aggregation Inhibition After a Single Subcutaneous Injection of ACT-246475 in Adults With Acute Myocardial Infarction
Brief Title: A Medical Research Study to Evaluate the Effects of ACT-246475 in Adults With Heart Attack
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID-076A202; 2018-000765-36 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-04-04 (Actual); Results first posted 2021-08-25 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2022-11

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — selatogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selatogrel 8 mg (Experimental): Selatogrel (ACT-246475) is given as a single subcutaneous dose of 8 mg administered in a volume of 0.8 mL. Administration will be performed at the investigational site by qualified personnel.
  Interventions: Drug: Selatogrel 8 mg
- Selatogrel 16 mg (Experimental): Selatogrel (ACT-246475) is given as a single subcutaneous dose of 16 mg administered in a volume of 0.8 mL. Administration will be performed at the investigational site by qualified personnel.
  Interventions: Drug: Selatogrel 16 mg

INTERVENTIONS:
Drug: Selatogrel 8 mg — Selatogrel is a reversible P2Y12 receptor antagonist for subcutaneous administration. It is supplied in sealed glass vials at a strength of 20 mg. The vials with ACT-246475A (hydrochloride salt of ACT-246475) will be reconstituted with 1 mL of water and further diluted with 1 mL sodium chloride (NaCl) 0.9%.
  Other Names: ACT-246475
  Arms: Selatogrel 8 mg
Drug: Selatogrel 16 mg — Selatogrel is a reversible P2Y12 receptor antagonist for subcutaneous administration. It is supplied in sealed glass vials at a strength of 20 mg. The vials with ACT-246475A (hydrochloride salt of ACT-246475) will be reconstituted with 1 mL of water for injection.
  Other Names: ACT-246475
  Arms: Selatogrel 16 mg

SUMMARY:
The goal of this study is to find out how fast a drug called selatogrel (ACT-246475) can prevent platelets from binding together. This study will also help to find out more about the safety of this new drug. The drug selatogrel (ACT-246475) will be used in 2 different doses (8 mg or 16 mg) and will be administered in the thigh.

DETAILED DESCRIPTION:
This study is planned in patients presenting with Acute Myocardial Infarction (AMI) scheduled for an invasive strategy. Platelet activation and thrombus formation play a pivotal role in the pathophysiology of acute coronary syndrome. Early platelet inhibition has been shown to reduce the risk of recurrent events after a myocardial infarction.

The screening period starts when the participant provides informed consent and ends with participant's randomization. Eligible participants had an acute myocardial infarction (AMI; ST-segment elevation myocardial infarction [STEMI] or non-ST-elevation myocardial infarction [NSTEMI]), a life-threatening condition, and will therefore fulfill the ICH-GCP definition of vulnerable subjects ("persons in emergency situations"). Accordingly, a specific process for obtaining consent in compliance with local regulations and approved by the independent ethics committee will be implemented.

The study will be performed during a participant's hospital stay related to the qualifying AMI.

Standard treatment of AMI is allowed including anticoagulants. Ticagrelor will be the only oral P2Y12 receptor antagonist allowed to be initiated during the study and its administration will be possible only after selatogrel administration. Use of fibrinolytics or GPIIb/IIIa inhibitors will be prohibited unless required for bail-out. All other standard-of-care treatments for AMI will be allowed without restriction.

The treatment period starts with the participant's randomization and ends after the end-of-study assessments, approximately 48 hours after the administration of a single study treatment dose.

ELIGIBILITY:
Main Inclusion Criteria:

* Informed consent obtained prior to any study-mandated procedure,
* Males aged from 18 to 85 and postmenopausal females aged up to 85 years,
* Onset of symptoms of AMI of more than 30 min and less than 6 hours prior to randomization,
* Subjects presenting a type I AMI including STEMI or NSTEMI.

Main Exclusion Criteria:

* Cardiogenic shock or severe hemodynamic instability,
* Cardiopulmonary resuscitation,
* Loading dose of any oral P2Y12 receptor antagonist prior to randomization,
* Planned fibrinolytic therapy or any fibrinolytic therapy administered within 24 h prior to randomization,
* Known platelet disorders (e.g., thromboasthenia, thrombocytopenia, von Willebrand disease).
* Active internal bleeding, or bleeding diathesis or conditions associated with high risk of bleeding.
* Known clinically important anemia.
* Oral anticoagulation therapy within 7 days prior to randomization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (6):
- Belgium (2):
  - OLV Ziekenhuis Aalst, Aalst
  - UZLeuven, Leuven
- Galilee Medical Center, Nahariya, Israel
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - University Hospital Bern, Bern
  - Cardiocentro Ticino, Lugano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurbel PA, Bliden KP, Butler K, Antonino MJ, Wei C, Teng R, Rasmussen L, Storey RF, Nielsen T, Eikelboom JW, Sabe-Affaki G, Husted S, Kereiakes DJ, Henderson D, Patel DV, Tantry US. Response to ticagrelor in clopidogrel nonresponders and responders and effect of switching therapies: the RESPOND study. Circulation. 2010 Mar 16;121(10):1188-99. doi: 10.1161/CIRCULATIONAHA.109.919456. Epub 2010 Mar 1. PMID 20194878
- [Background] Jernberg T, Payne CD, Winters KJ, Darstein C, Brandt JT, Jakubowski JA, Naganuma H, Siegbahn A, Wallentin L. Prasugrel achieves greater inhibition of platelet aggregation and a lower rate of non-responders compared with clopidogrel in aspirin-treated patients with stable coronary artery disease. Eur Heart J. 2006 May;27(10):1166-73. doi: 10.1093/eurheartj/ehi877. Epub 2006 Apr 18. PMID 16621870
- [Background] Parodi G, Bellandi B, Valenti R, Migliorini A, Marcucci R, Carrabba N, Giurlani L, Gensini GF, Abbate R, Antoniucci D. Comparison of double (360 mg) ticagrelor loading dose with standard (60 mg) prasugrel loading dose in ST-elevation myocardial infarction patients: the Rapid Activity of Platelet Inhibitor Drugs (RAPID) primary PCI 2 study. Am Heart J. 2014 Jun;167(6):909-14. doi: 10.1016/j.ahj.2014.03.011. Epub 2014 Apr 4. PMID 24890542
- [Derived] Sinnaeve P, Fahrni G, Schelfaut D, Spirito A, Mueller C, Frenoux JM, Hmissi A, Bernaud C, Ufer M, Moccetti T, Atar S, Valgimigli M. Subcutaneous Selatogrel Inhibits Platelet Aggregation in Patients With Acute Myocardial Infarction. J Am Coll Cardiol. 2020 May 26;75(20):2588-2597. doi: 10.1016/j.jacc.2020.03.059. PMID 32439008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 10 July and 10 November 2018. Seven sites were initiated. Six sites in 3 countries screened and randomized 48 participants.
Pre-assignment Details: Forty-eight patients were randomized to either selatogrel 8 mg or 16 mg. Forty-seven patients were administered selatogrel and completed the study. One patient randomized to the 8 mg group did not receive selatogrel (not treated for administrative reasons) and was excluded from the full-analysis set (FAS).
Groups:
- Selatogrel 8 mg: A single 8 mg dose of selatogrel (ACT-246475) was administered via a single subcutaneous injection in the thigh.
- Selatogrel 16 mg: A single 16 mg dose of selatogrel (ACT-246475) was administered via a single subcutaneous injection in the thigh.
Period: Randomization
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Started | 25 | 23
Completed | 24 | 23
Not Completed | 1 | 0
Not completed — Not treated for administrative reasons | 1 | 0
Period: Treatment Period
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Started | 24 | 23
Modified Full Analysis Set (mFAS) (mFAS: all participants with a 30-min post dose VerifyNow® blood sample analysis.) | 23 | 22
Per Protocol Set | 20 | 20
Completed | 24 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (all participants that were treated).
Groups:
- Total: Total of all reporting groups
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants] — Population: The per-protocol set includes all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  Participants
    Full Analysis Set: <=18 years | 0 | 0 | 0
    Full Analysis Set: Between 18 and 65 years | 9 | 8 | 17
    Full Analysis Set: >=65 years | 15 | 15 | 30
    Per Protocol Set: number analyzed (Participants) | 20 | 20 | 40
    Per Protocol Set: <=18 years | 0 | 0 | 0
    Per Protocol Set: Between 18 and 65 years | 9 | 7 | 16
    Per Protocol Set: >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The per-protocol set includes all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  years
    Full Analysis Set | 65.5 (11.3) | 68.0 (10.3) | 66.7 (10.8)
    Per Protocol Set: number analyzed (Participants) | 20 | 20 | 40
    Per Protocol Set | 64.5 (12.1) | 67.9 (10.3) | 66.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The per-protocol set includes all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  Participants
    Full Analysis Set: Female | 8 | 5 | 13
    Full Analysis Set: Male | 16 | 18 | 34
    Per Protocol Set: number analyzed (Participants) | 20 | 20 | 40
    Per Protocol Set: Female | 5 | 4 | 9
    Per Protocol Set: Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The per-protocol set includes all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  Participants
    Full Analysis Set: Hispanic or Latino | 0 | 0 | 0
    Full Analysis Set: Not Hispanic or Latino | 24 | 23 | 47
    Full Analysis Set: Unknown or Not Reported | 0 | 0 | 0
    Per Protocol Set: number analyzed (Participants) | 20 | 20 | 40
    Per Protocol Set: Hispanic or Latino | 0 | 0 | 0
    Per Protocol Set: Not Hispanic or Latino | 20 | 20 | 40
    Per Protocol Set: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The per-protocol set includes all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  Participants
    Full Analysis Set: American Indian or Alaska Native | 0 | 0 | 0
    Full Analysis Set: Asian | 1 | 2 | 3
    Full Analysis Set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Full Analysis Set: Black or African American | 0 | 0 | 0
    Full Analysis Set: White | 22 | 21 | 43
    Full Analysis Set: More than one race | 0 | 0 | 0
    Full Analysis Set: Unknown or Not Reported | 1 | 0 | 1
    Per Protocol Set: number analyzed (Participants) | 20 | 20 | 40
    Per Protocol Set: American Indian or Alaska Native | 0 | 0 | 0
    Per Protocol Set: Asian | 1 | 2 | 3
    Per Protocol Set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Per Protocol Set: Black or African American | 0 | 0 | 0
    Per Protocol Set: White | 18 | 18 | 36
    Per Protocol Set: More than one race | 0 | 0 | 0
    Per Protocol Set: Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 7 | 7 | 14
  Israel | 1 | 0 | 1
  Switzerland | 16 | 16 | 32
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] — at screening visit
  kilograms per square meter
    Full Analysis Set | 28.00 (4.83) | 26.78 (3.74) | 27.40 (4.33)
    Per Protocol Set | 27.64 (4.88) | 26.67 (3.79) | 27.16 (4.34)
Medical history risk factors at baseline [Count of Participants; unit: Participants]
  Diabetes mellitus | 8 | 5 | 13
  Chronic Kidney disease | 0 | 3 | 3
  Hypertension | 15 | 12 | 27
  Dyslipidemia | 8 | 10 | 18
Diagnosis at enrollment [Count of Participants; unit: Participants] — Eligible participants presented with acute myocardial infarction (STEMI [ST-segment elevation myocardial infarction] or NSTEMI [Non-ST-segment elevation myocardial infarction]).
  Participants
    NSTEMI | 8 | 10 | 18
    STEMI | 16 | 13 | 29
STEMI: Thrombolysis in myocardial infarction (TIMI) risk score [Count of Participants; unit: Participants] — The TIMI score is used to make clinical decisions about patient management and predicting the likelihood of adverse cardiac events. In STEMI participants the score ranges from 0 to 14. A higher TIMI score indicates a higher risk of adverse cardiac events. TIMI scores below 3 constitute a low risk of cardiac adverse events in the next month. TIMI scores of 3 and above constitute a moderate to high risk. Population: Participants diagnosis at enrollment with STEMI (ST-segment elevation myocardial infarction)
  Participants
    number analyzed (Participants) | 16 | 13 | 29
    STEMI : TIMI Risk Score less than 3 | 9 | 6 | 15
    STEMI : TIMI Risk Score 3 or greater | 7 | 7 | 14
NSTEMI: Thrombolysis in myocardial infarction (TIMI) risk score [Count of Participants; unit: Participants] — The TIMI score is used to make clinical decisions about patient management and predicting the likelihood of adverse cardiac events. In NSTEMI participants scores range from 0 to 7. A higher TIMI score indicates a higher risk of adverse cardiac events. Scores of less than 5 constitutes a low risk of adverse cardiac events in the next 14 days and scores of 5 and above constitute a moderate to high risk. Population: Participants diagnosis at enrollment with NSTEMI (Non-ST-segment elevation myocardial infarction)
  Participants
    number analyzed (Participants) | 8 | 10 | 18
    NSTEMI: TIMI risk score less than 5 | 6 | 6 | 12
    NSTEMI: TIMI risk score 5 and above | 2 | 4 | 6
Time from onset of acute myocardial infarction symptoms to treatment start [Mean (Standard Deviation); unit: hours] | 4.00 (1.64) | 3.85 (1.56) | 3.93 (1.59)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Pharmacodynamic Response as Assessed by the Inhibition of Platelet Aggregation
Description: The pharmacodynamic response was determined by measuring the inhibition of platelet aggregation, using the VerifyNow® assay. The VerifyNow® is a point-of-care test measuring platelet reactivity. The results are expressed as P2Y12 reaction units (PRU).The target of 100 PRU corresponds to 80% inhibition of ADP-induced platelet aggregation. A participant with a PRU less than 100 at 30 minutes post-dose was counted as a participant that had a pharmacodynamic response.
Time Frame: 30 minutes after the administration of the subcutaneous injection
Population: The modified full analysis set (mFAS) includes all participants from the FAS who have an assessment of the primary endpoint (that is all participants with a 30-min post dose VerifyNow® blood sample analysis).
Measure: Number; unit: Count of participants
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 23 | 22
Count of participants | 21 | 21
Statistical Analysis 1: Comparison: Selatogrel 8 mg; The main analysis (mFAS, treatment dose as received) of treatment effect on the primary endpoint was conducted independently for each dose; Test type: Superiority — The statistical analysis comprised a 2-step testing strategy. The first test, carried out at an alpha level of 0.025, determined whether the proportion of responders (patients with a PRU value <100) was ≥ 50% (null hypothesis: proportion of responders <50%) and is reported below. The second step for the Selatogrel 8 mg is described in statistical analysis 2: In this second analysis the subsequent null hypothesis of treatment effect less or equal to 85% was tested for the 8 mg dose; p < 0.001, one-sided z-test — P-value for hypotheses (H0: p <= 50% vs. H1: p > 50%); A p-value significance level was set to 0.025
Statistical Analysis 2: Comparison: Selatogrel 8 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This statistical analysis reports the second of the 2-step testing strategy. This second test for the 8 mg Selatogrel dose, carried out at an alpha level of 0.025, determined whether the proportion of responders (patients with a PRU value <100) was ≥ 85% (null hypothesis: proportion of responders <85%); p = 0.142, one-sided z-test — P-value for hypotheses (H0: p <= 85% vs. H1: p > 85%); A p-value significance level was set to 0.025, an overall level of 0.05 and adjusted for multiplicity using the Bonferroni approach
Statistical Analysis 3: Comparison: Selatogrel 16 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The statistical analysis comprised a 2-step testing strategy. The first test, carried out at an alpha level of 0.025, determined whether the proportion of responders (patients with a PRU value <100) was ≥ 50% (null hypothesis: proportion of responders <50%) and is reported below. The second step for the Selatogrel 16 mg is described in statistical analysis 4: In this second analysis the subsequent null hypothesis of treatment effect less or equal to 85% was tested for the 16 mg dose; p < 0.0001, one-sided z-test — P-value for hypotheses (H0: p <= 50% vs. H1: p > 50%); A p-value significance level was set to 0.025
Statistical Analysis 4: Comparison: Selatogrel 16 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — This statistical analysis reports the second of the 2-step testing strategy. This second test for the 16 mg Selatogrel dose, carried out at an alpha level of 0.025, determined whether the proportion of responders (patients with a PRU value <100) was ≥ 85% (null hypothesis: proportion of responders <85%); p = 0.009, one-sided z-test — P-value for hypotheses (H0: p <= 85% vs. H1: p > 85%); [statistical method as in outcome 1, analysis 2]

2. Other Pre Specified Outcome: Number of Participants (Per-protocol Subgroup) With a Pharmacodynamic Response as Assessed by the Inhibition of Platelet Aggregation
Description: The pharmacodynamic response was determined by measuring the inhibition of platelet aggregation, using VerifyNow®. The VerifyNow® is a point-of-care test measuring platelet reactivity. The results are expressed as P2Y12 reaction units (PRU). The target of 100 PRU corresponds to 80% inhibition of ADP-induced platelet aggregation. A participant with a PRU of less than 100 starting at 30 minutes post-dose was counted as a participant that had a pharmacodynamic response.
Time Frame: 30 minutes after the administration of the subcutaneous injection
Population: Supportive analysis of the primary endpoint: per-protocol set
Measure: Number; unit: Count of participants
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 20 | 20
Count of participants | 18 | 19
Statistical Analysis 1: Comparison: Selatogrel 8 mg; As per the main analysis (mFAS) the supporting analysis on the per-protocol set this analysis of treatment effect was conducted independently for each dose, i.e., 8 and 16 mg; Test type: Superiority; p = 0.2280, One-sided Z-test — P-value for hypotheses (H0: p <= 85% versus H1: p > 85%)
Statistical Analysis 2: Comparison: Selatogrel 16 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0201, One-sided Z-test — P-value for hypotheses (H0: p <= 85% versus H1: p > 85%)

3. Other Pre Specified Outcome: Number of Participants With a Pharmacodynamic Response Within the First Hour as Assessed by the Inhibition of Platelet Aggregation
Description: The purpose of this supportive analysis was to assess the effect when relaxing the time of a PRU < 100, i.e., considering as a response a PRU < 100 at 15, 30 or 60 min. post injection. The pharmacodynamic response was determined by measuring the inhibition of platelet aggregation, using the VerifyNow® assay. The VerifyNow® is a point-of-care test measuring platelet reactivity. The results are expressed as P2Y12 reaction units (PRU).The target of 100 PRU corresponds to 80% inhibition of ADP-induced platelet aggregation. A participant with a PRU less than 100 post-dose was counted as a participant that had a pharmacodynamic response.
Time Frame: pre-dose, 15, 30 and 60 minutes after the administration of the subcutaneous injection
Population: Full analysis set
Measure: Number; unit: Count of participants
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 24 | 23
Count of participants
  pre-dose | 1 | 0
  15 minutes post-dose | 18 | 21
  30 minutes post-dose | 21 | 21
  60 minutes post-dose | 18 | 22

4. Other Pre Specified Outcome: Absolute Platelet Reactivity (P2Y12 Reaction Units) Over Time
Description: The pharmacodynamic response assessed by the inhibition of adenosine diphosphate (ADP)-mediated platelet aggregation was determined by measuring the inhibition of platelet aggregation, using VerifyNow®. The VerifyNow® is a point-of-care test. The results are expressed as P2Y12 reaction units (PRU).
Time Frame: pre-dose, 15, 30 and 60 minutes after administration of the subcutaneous injection
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: P2Y12 reaction units (PRU)
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 24 | 23
P2Y12 reaction units (PRU)
  pre-dose | 194 [159 to 213] | 181 [148 to 213]
  15 minutes post-dose | 51 [4 to 208] | 9 [2 to 282]
  30 minutes post-dose | 59 [2 to 135] | 9 [2 to 117]
  60 minutes post-dose | 9 [2 to 116] | 7 [1 to 228]

5. Other Pre Specified Outcome: Maximum Selatogrel Plasma Concentration (Cmax)
Description: The Cmax is the peak concentration of selatogrel in the plasma after subcutaneous injection.
  The pharmacokinetic parameters of selatogrel (ACT-246475) were derived by non-compartmental analyses of the plasma concentration-time profiles.
Time Frame: pre-dose, 15, 30 and 60 minutes and 8 hours after the administration of the subcutaneous injection
Population: Pharmacokinetic analysis set - all participants that had at least one selatogrel concentration measurement after administration of study treatment.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 24 | 22
ng/mL | 390.1 [206 to 848] | 672.6 [276 to 1180]

6. Other Pre Specified Outcome: Time to Reach Maximum Selatogrel Plasma Concentration (Tmax)
Description: Time after subcutaneous injection to reach the maximum observed selatogrel plasma concentration (Cmax).
Time Frame: pre-dose, 15, 30 and 60 minutes and 8 hours after the administration of the subcutaneous injection
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 24 | 22
hours | 1.00 [0.50 to 1.27] | 0.97 [0.25 to 1.15]

7. Post Hoc Outcome: Subgroup Analyses: Number of Participants With a Pharmacodynamic Response as Assessed by the Inhibition of Platelet Aggregation
Description: as for outcome 2
Time Frame: 30 minutes after the administration of the subcutaneous injection
Population: Full Analysis Set
Measure: Number; unit: Count of participants
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 24 | 23
Count of participants
  Age less than 55 years old: number analyzed (Participants) | 4 | 4
  Age less than 55 years old | 3 | 4
  Age 55 years and older: number analyzed (Participants) | 20 | 19
  Age 55 years and older | 18 | 17
  Male: number analyzed (Participants) | 16 | 18
  Male | 14 | 17
  Female: number analyzed (Participants) | 8 | 5
  Female | 7 | 4
  Body Mass Index less than 25: number analyzed (Participants) | 7 | 9
  Body Mass Index less than 25 | 5 | 8
  Body Mass Index less than 25 and up to 30: number analyzed (Participants) | 8 | 10
  Body Mass Index less than 25 and up to 30 | 8 | 9
  Body Mass Index greater than 30: number analyzed (Participants) | 9 | 4
  Body Mass Index greater than 30 | 8 | 4
  Diabetes mellitus at baseline: number analyzed (Participants) | 8 | 5
  Diabetes mellitus at baseline | 8 | 5
  No diabetes mellitus at baseline: number analyzed (Participants) | 16 | 18
  No diabetes mellitus at baseline | 13 | 16
  Chronic kidney disease at baseline: number analyzed (Participants) | 0 | 3
  Chronic kidney disease at baseline |  | 3
  No Chronic kidney disease at baseline: number analyzed (Participants) | 24 | 20
  No Chronic kidney disease at baseline | 21 | 18
  STEMI at baseline: number analyzed (Participants) | 16 | 13
  STEMI at baseline | 14 | 11
  NSTEMI at baseline: number analyzed (Participants) | 8 | 10
  NSTEMI at baseline | 7 | 10

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were those adverse events with onset after study drug administration and up to 48 hours after study treatment administration.
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/23
Other Adverse Events (participants affected / at risk) | 12/24 | 7/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selatogrel 8 mg (N=24) | Selatogrel 16 mg (N=23)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selatogrel 8 mg (N=24) | Selatogrel 16 mg (N=23)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The p-values need to be cautiously interpreted due to the small study population size.

The participants were expected per protocol to shortly undergo invasive management, it was anticipated that most would receive an early loading dose of ticagrelor.

Blood samples were collected with phenylalanine-proline-arginine-chloromethylketone as anticoagulant.

Only the VerifyNow® assay was used to assess the platelet response to selatogrel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03487445/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT03487445/SAP_001.pdf